CLINICAL TRIAL: NCT01840176
Title: Prophylactic Modified McCall Culdoplasty During Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 13-0101
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Vaginal Vault Prolapse; Sexual Function
Keywords: McCall culdoplasty; Total laparoscopic hysterectomy; Vaginal vault prolapse; Sexual function
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine (No Intervention): These women are randomized to receive no McCall culdoplasty at the time of their total laparoscopic hysterectomy.
- McCall culdoplasty (Other): The women in this arm are those randomized to undergo a McCall culdoplasty at the time of their total laparoscopic hysterectomy.
  Interventions: Procedure: McCall culdoplasty

INTERVENTIONS:
Procedure: McCall culdoplasty — The modified McCall Culdoplasty procedure is a relatively simple procedure that is performed after removal of the uterus and cervix from the apex of the vagina wherein the angles of the vagina are attached to their respective uterosacral ligament and the cul-de-sac is surgically obliterated for support postoperatively. This is done with a single 0-vicryl suture. There will be no additional interventions applied during the hysterectomy aside from the McCall culdoplasty.
  Arms: McCall culdoplasty

SUMMARY:
The purpose of this study is to assess the feasibility of performing prophylactic McCall culdoplasty at the time of total laparoscopic hysterectomy. The investigators will also be measuring pelvic support (using POP-Q) and sexual function before and at different time points (up to 12 months) postoperatively.

The investigators hypothesize that women undergoing the McCall culdoplasty will not have different immediate surgical outcomes (operative time, etc) and may have better pelvic support and sexual function in the future.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-99 undergoing elective laparoscopic hysterectomy for benign indications with surgeons in the division of Advanced Laparoscopy and Pelvic Pain at UNC-Chapel Hill.

Exclusion Criteria:

* Current symptomatic or asymptomatic pelvic organ prolapse as measured by the Pelvic Organ Prolapse Quantification (POPQ) system.
* Pregnancy
* Non-English speaking
* Unable to provide informed consent
* Pathology causing an obliterated cul-de-sac

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | 6 months
  The primary aim of the study is to generate feasibility data for performing a powered randomized trial on prophylactic modified McCall's culdoplasty during benign total laparoscopic hysterectomy. As such, we will measure operative time with the hypothesis that the intervention does not add significant additional effort. We will also collect information regarding patient willingness to participate as well as intra- and post-operative complication data.

SECONDARY OUTCOMES:
Pelvic support | 12 months
  This study will also allow us to collect data regarding differences in POP-Q exams up to 12 months after surgery.
Sexual function | 12 months
  We will also collect data regarding sexual function at different time points pre and postoperatively up to 12 months after surgery using the validated Female Sexual Function Index (FSFI) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kumari Hobbs, MD, Principal Investigator — UNC Chapel Hill Dept of OB/GYN; Matthew Siedhoff, MD, Study Director — UNC Chapel Hill Dept of OB/GYN
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Till SR, Hobbs KA, Moulder JK, Steege JF, Siedhoff MT. McCall Culdoplasty during Total Laparoscopic Hysterectomy: A Pilot Randomized Controlled Trial. J Minim Invasive Gynecol. 2018 May-Jun;25(4):670-678. doi: 10.1016/j.jmig.2017.10.036. Epub 2017 Nov 8. PMID 29128440